## **Informed Consent**

NCT05708846

5th May 2023

## **Participant Consent:**

| , | <del></del> |
|---|---|
| improvement of a digital health platform fo | been given to me about the "Observational study for the remote monitoring of patients with heart failure", with ter Followhealth S.L., the "study" from now on: |
| - I am aware that the data collected will be | used solely for the purposes of the "study" and that the |
| minimum data necessary to achieve its object | ctives will be collected. |
| also been informed of who the responsible | ives of the "study" for which the data is collected. I have team is and I have been given contact information with the information collected and/or to request access to my |
| - I know that the data will be stored on a sec | ure server. |
| appropriate to me, I understand the risk participation in it is voluntary and that I can I understand that the "study" information | had the opportunity to ask the questions that seemed<br>s and benefits that arise from the study and that my<br>withdraw from it at any time.<br>will be confidential and that no unauthorized person will |
| have access to the data. | , from |
| - I know how to contact the doctor if I need t | |
| - I have received enough information about t | |
| - I understand that I can withdraw from the ' | |
| | study . |
| - Whenever I want. | |
| - Without having to explain. | |
| - Without this affecting my medical care. | |
| the Council of April 26, 2016 regarding the processing of personal data, the purpose in accordance with the provisions of arts. Securopean Parliament and of the Council, of 3/2018, of December 5, Protection of Personal data, the purpose in accordance with the provisions of arts. | ulation EU 2016/679 of the European Parliament and of rotection of natural persons in terms of the processing of ta, I declare that I have been informed of the existence of e of collecting them and the recipients of the information 5, 6, 7, 12 and/or 13 of Regulation (EU) 2016/679 of the April 27, 2016 (RGPD) as well as in art. 11 of Organic Lawnal Data and guarantee of digital rights (LOPD). |
| - I freely give my consent to participate in the | e study. |
| Signature of the participant | Physician Signature |
| Date:/ D. | ate:/ |

| Revoc | ation of consent | <u>:</u> | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| The | undersigned | patient | revokes | the | consent | granted | to | doctor | Dr |
| | | | | for his p | articipation | in the " <i>Obse</i> | ervatio | nal study fo | or the |
| impro | vement of a digit | al health pl | atform for t | he remo | te monitorin | g of patients | with h | eart failure | ?". |
| Signature of the participant | | | | Physician Signature | | | | | |
| Date: | / | | Dat | te:/ | '/_ | | | | |